CLINICAL TRIAL: NCT06347770
Title: Effect of Probiotics Before Cesarean Section on Postoperative Recovery in Pregnant Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhe Li, Principal Investigator, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ThirdSunYat-senECII202329903
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Microbiota; Postoperative Recovery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): pregnancies in control group need no intervention
- probiotics group (Experimental): pregnancies in probiotics group need probiotics management
  Interventions: Drug: Probiotic Blend Oral Tablet

INTERVENTIONS:
Drug: Probiotic Blend Oral Tablet — In our study, forty pregnant women were randomly assigned to the probiotic group, and the rest were assigned to the control group. After enrollment, pregnant women in the probiotic group received a combination of living Bifidobacterium longum (5 #106 CFU) by Neimengu Shuangqi Pharmaceutical Co., Ltd. Pregnant individuals in the probiotic group were administered four tablets three times a day (2 g/d) for seven days before surgery until the fourth day after surgery.
  Arms: probiotics group

SUMMARY:
This study aims to evaluate the effect of probiotics 7 days before cesarean section (CS) on postoperative recovery and the change of gut microbiota in pregnant women. Samples were obtained from a total of 80 pregnant individuals, divided into control group and probiotics group. Anal exhaust time and first defecating time were set as the primary outcome of recovery of CS. 16S rRNA amplicon sequencing of the V4 region was analyzed to evaluate the composition of them.

DETAILED DESCRIPTION:
Study design and participants A total of 80 samples were obtained from pregnant individuals receiving antenatal care at the 3rd Affiliated Hospital of Sun Yat-sen University and the 1st Affiliated Hospital of Jinan University. Informed consent was obtained from pregnant women (at least 32 gestational weeks) who met the inclusion criteria. Pregnant women were followed until 7 days after cesarean section. Pregnant inclusive criteria were: 1. Chinese woman who is pregnant with a single fetus; 2. Pregnant women who planned to perform lower section of uterus due to social factors, relative head basin asymmetry, macrosomia, cicatricial uterus and other reasons. Pregnant exclusive criteria were: 1. Gastrointestinal disease or family history; 2. Antibiotic usage during pregnancy; 3. Habit of eating foods with high probiotic content such as yogurt and cheese during pregnancy; 4. Take other probiotics or probiotic drinks during pregnancy regularly; 5. Hypertension, Diabetes Mellitus, Hyperthyroidism, Hypothyroidism, Autoimmune Disease, or Other Endocrine and Metabolic Disease; 6. Transfusion History, Organ Transplantation History or Immunotherapy; 7. Gestational hypertension, gestational diabetes, gestational thyroid dysfunction and other endocrine and metabolic diseases occurred during this pregnancy.

Probiotic management In our study, forty pregnant women were randomly assigned to the probiotic group, and the rest were assigned to the control group. After enrollment, pregnant women in the probiotic group received the living Bifidobacterium longum (5 # 106 CFU) tablets produced by Neimengu Shuangqi Pharmaceutical Co., Ltd. Pregnant individuals in the probiotic group were administered four tablets three times a day (2 g/d) for seven days before surgery until the fourth day after surgery, and those in the control group took no pills.

Fecal, venous blood and data collection Fecal collection Feces from pregnant women were collected twice-the last time before surgery and the first time after surgery. Feces collected were both collected internally, thereby avoiding contamination with foreign material. The feces were transferred to the laboratory freezer at 80ºC within 30 min of collection when obtained in the hospital. Feces collected were stored in a domestic refrigerator and transferred to the laboratory freezer for 24 hours when obtained outside the hospital.

Venous blood collection Venous blood from pregnant women was collected twice-before and after surgery. The venous blood was obtained in the hospital and centrifuged within 30 minutes in a temperature-controlled centrifuge at 3000 r/min at 4℃ for 10 minutes after 2ml of which was collected, then the serum samples were transferred to the laboratory freezer at -80ºC.

Data collection Data from pregnant women was collected before and after surgery, including age, height, pre-delivery weight, time of first anal exhaust and defecation.

ELIGIBILITY:
Inclusion Criteria:

* Chinese woman who is pregnant with a single fetus
* Pregnant women who planned to perform lower section of uterus due to social factors, relative head basin asymmetry, macrosomia, cicatricial uterus and other reasons.

Exclusion Criteria:

* Gastrointestinal disease or family history
* Antibiotic usage during pregnancy
* Habit of eating foods with high probiotic content such as yogurt and cheese during pregnancy
* Take other probiotics or probiotic drinks during pregnancy regularly
* Hypertension, Diabetes Mellitus, Hyperthyroidism, Hypothyroidism, Autoimmune Disease, or Other Endocrine and Metabolic Disease
* Transfusion History, Organ Transplantation History or Immunotherapy
* Gestational hypertension, gestational diabetes, gestational thyroid dysfunction and other endocrine and metabolic diseases occurred during this pregnancy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
analysis of postoperative recovery | 12 months
  The specific time between the first postoperative exhaust, defecation and the completion of the operation as well as the outcome of blood routine examination were collected. Difference analysis of each group was performed. All the measurement data are presented as the mean ± standard error. Assessments of Operational Taxonomic Units differences in the probiotic group and control group were performed using independent sample t tests, and P < 0.05 was considered to indicate statistical significance. Other outcomes were analyzed using multiple linear regression. All data were analyzed using SPSS 23.0 statistical software (SPSS, Inc., Chicago, IL, USA).
16S rRNA amplicon sequencing of the V4 region | 12 months
  Difference analysis of each group was performed. All the measurement data are presented as the mean ± standard error. Assessments of Operational Taxonomic Units differences in the probiotic group and control group were performed using independent sample t tests, and P < 0.05 was considered to indicate statistical significance. Other outcomes were analyzed using multiple linear regression. All data were analyzed using SPSS 23.0 statistical software (SPSS, Inc., Chicago, IL, USA).

CONTACTS AND LOCATIONS:
Locations (1):
- Zhe Li, Guangzhou, Guangdong, China